CLINICAL TRIAL: NCT01333917
Title: Curcumin Chemoprevention of Colorectal Neoplasia
Brief Title: Curcumin Biomarkers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 10-1524
Record Dates: First submitted 2011-04-06; First posted 2011-04-12 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer
Keywords: Curcumin; Colorectal Cancer; GWAS
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Curcumin (Experimental): 4g Curcumin C3 tablet daily
  Interventions: Drug: Curcumin C3 tablet

INTERVENTIONS:
Drug: Curcumin C3 tablet — 4 grams Curcumin C3 tablet daily x30 days

SUMMARY:
Colorectal cancer is a major problem in the United States and other developed countries. A safe and effective chemopreventive agent could reduce the burden of colorectal neoplasia. Curcumin, is a product that is derived from Curcuma longa. It has been used for thousands of years as a traditional remedy. Curcumin blocks a number of targets involved in tumor initiation, promotion, and progression, and is considered a promising chemopreventive agent. The investigators propose to enroll 40 patients after screening colonoscopy who will have rectal biopsies at baseline and after 4 weeks of curcumin 4 grams per day. The investigators will use microarray analysis to identify genes that are modified by curcumin that could be used as biomarkers in future chemoprevention studies. The study will also evaluate tolerability and toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 - 80.
2. A willingness to follow the study protocol, as indicated by provision of informed consent to participate
3. Good general health

Exclusion Criteria:

1. Familial colorectal cancer syndromes (e.g. Hereditary Non-Polyposis Colon Cancer, Familial Adenomatous Polyposis)
2. Ulcerative colitis or Crohn's disease.
3. History of large bowel resection for any reason
4. Diagnosed narcotic or alcohol dependence
5. Unwillingness to forgo curcumin/turmeric-containing supplements during the trial or consumption of curry/turmeric at meals > 3 times a week.
6. Allergy to turmeric/curcumin.
7. Women with childbearing potential who do not agree to practice effective birth control.
8. Individuals with creatinine, AST or ALT above 1.5 times the upper limit of normal at baseline.
9. Personal or inherited bleeding disorders or therapeutic anti-coagulation with warfarin.
10. Women who are pregnant or nursing.
11. Individuals who have taken antibiotics within the three months prior to enrollment.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Gene expression | 30 days
  Change in gene expression
Ribonucleic acid (RNA) level | 30 days
  Transcript level as mRNA copies per cell
Apoptosis | 30 days
  Immunohistochemistry (IHC) signal as intensity and proportion of cells stained

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Gary N Asher, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Department of Family Medicine, Chapel Hill, North Carolina, United States